CLINICAL TRIAL: NCT03392896
Title: A Placebo-Controlled, Single-Blind, Single-Center Phase 1 Study in Normal Healthy Volunteers and Open-Label Multi-Center Study in Patients With Primary Hyperoxaluria to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Doses of DCR-PHXC Solution for Injection (Subcutaneous Use)
Brief Title: Study of DCR-PHXC-101 in Normal Healthy Volunteers and Patients With Primary Hyperoxaluria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dicerna Pharmaceuticals, Inc., a Novo Nordisk company (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DCR-PHXC-101
Record Dates: First submitted 2017-12-21; First posted 2018-01-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Primary Hyperoxaluria
MeSH Terms: conditions — Hyperoxaluria, Primary

STUDY DESIGN:
Intervention Model Description: Two-arm (active and placebo), single-blind, SAD period (Group A, HVs) followed by open-label, SAD period (Group B, PH1 and PH2 patients).
Who Masked: Participant, Investigator
Masking Description: SAD period in HV is single-blind (unblinded clinical site staff member who is not a member of study team administers dose). SAD period in Group B (PH1 and PH2 patients) is open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group A Active (DCR-PHXC) (Experimental): HVs, single ascending doses of DCR-PHXC.
  Interventions: Drug: DCR-PHXC
- Group A Placebo (Placebo Comparator): HVs, normal saline 0.9% injection to match active doses.
  Interventions: Drug: Placebo
- Group B Active (DCR-PHXC) (Experimental): PH1 and PH2 patients, open label, single ascending doses of DCR-PHXC.
  Interventions: Drug: DCR-PHXC

INTERVENTIONS:
Drug: DCR-PHXC — DCR-PHXC is a novel, potent, and long-acting small interference ribonucleic acid (siRNA) molecule conjugated to N-acteylgalactosamine (GalNAc) that is designed to decrease liver oxalate production. DCR-PHXC is delivered via subcutaneous (SC) injection.
  Arms: Group A Active (DCR-PHXC); Group B Active (DCR-PHXC)
Drug: Placebo — Single SC administration of placebo, which will be a sterile, preservative-free normal saline 0.9% solution for SC injection, which is of similar osmolality to the DCR-PHXC formulation.
  Arms: Group A Placebo

SUMMARY:
This is a double-blind, placebo-controlled, dose escalation trial of DCR-PHXC in Healthy Volunteers (HVs) and patients with Primary Hyperoxaluria (PH). Once safety has been established in HV, PH patients with a confirmed diagnosis of PH1 and PH2 will be enrolled across multiple dosing cohorts. The study design will allow enrollment of PH patient cohorts at a given dose level once safety has been demonstrated in HV at that dose level. The study will be conducted in two parts: Part A: Single ascending dose (SAD) in HV; Part B: SAD in patients with PH1 and PH2 (lagging Part A by 1 dose level cohort).

ELIGIBILITY:
Group A (HVs) Major Inclusion Criteria:

* Willing and able to provide informed consent and comply with study requirements.
* Male or female subjects between 18 and 55 years of age, inclusive.
* Subject must have a body mass index (BMI) 19.0 to 32 kg/m2, inclusive.
* Non-smokers, at least 1-month tobacco free, and willing to remain tobacco free through end of study (EOS).
* Women of child bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be willing to use contraception.

Group A (HVs) Major Exclusion Criteria:

* Presence of any medical condition, including but not limited to: Severe intercurrent illness, known causes of active liver disease.
* Routine or chronic use of more than 3 grams of acetaminophen (Tylenol) daily.
* History of kidney stones.
* Use of any investigational agent within 90 days before the first dose of study medication.
* History of donation of more than 450 mL of blood within 90 days prior to dosing in the clinical research center or planned donation less than 30 days after receiving Investigational Medicinal Product (IMP).
* Plasma or platelet donation within 7 days of dosing and through EOS.
* History of reactions to an oligonucleotide-based therapy.
* Males with female partners who are planning to attempt to become pregnant during this study or within 90 days after last dosing of IMP.
* Plasma or platelet donation within 7 days of dosing and through EOS.

Group B (PH1 and PH2 patients) Major Inclusion Criteria:

* Willing and able to provide informed consent and comply with study requirements.
* Male or female, at least 6 years of age.
* Minimum body weight of 25 kg.
* Genetic confirmation of PH1 and PH2 disease.
* Meet the 24 hour urine oxalate excretion requirements.
* Estimated glomerular filtration rate (eGFR) ≥30 mL/min/1.73 m2.
* If taking Vitamin B6 (pyridoxine), must have been on stable regimen for at least 4 weeks.

Group B (PH1 and PH2 patients) Major Exclusion Criteria:

* Prior renal and/or hepatic transplantation.
* Currently receiving dialysis.
* Participation in any clinical study where they received an investigational agent within 4 months before enrollment.
* Presence of any medical condition, including but not limited to: Severe intercurrent illness, known causes of active liver disease.
* Liver function test (LFT) abnormalities.
* History of reactions to an oligonucleotide-based therapy.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-11-19 (Actual)

PRIMARY OUTCOMES:
Number of patients with Treatment-Related Adverse Events (TEAEs) | Part A (SAD in HVs) screening through Day 29; Part B (SAD in PH patients) screening through Day 57

CONTACTS AND LOCATIONS:
Locations (7):
- Boston Children's Hospital, Boston, Massachusetts, United States
- Centre d'Investigation Clinique - CIC 1407 - Hospices Civils de Lyon, Bron, France
- Universitätsklinikum Bonn-Institut für Klinische Chemie und Klinische Pharmakologie, Bonn, Germany
- University of Amsterdam, Amsterdam, Netherlands
- United Kingdom (3):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Birmingham Children's Hospital NHS Trust, Birmingham
  - Clinical Trial Site, Wales

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang S, Gamallo P, Rawson V. Population Pharmacokinetic and Pharmacodynamic Modelling and Simulation for Nedosiran Clinical Development and Dose Guidance in Pediatric Patients with Primary Hyperoxaluria Type 1. Clin Pharmacokinet. 2025 Sep;64(9):1395-1411. doi: 10.1007/s40262-025-01540-1. Epub 2025 Jul 2. PMID 40601241